CLINICAL TRIAL: NCT06025292
Title: Effects of Lean Pork Loin Intake on Protein Homeostasis and Glucose Regulation in Prediabetic Adults
Acronym: PORK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Pork Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 276210
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hyperglycaemia (Non Diabetic); Prediabetes
Keywords: Lean pork; Muscle Protein Synthesis; Protein; Plant-Based
MeSH Terms: conditions — Hyperglycemia; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Quality Protein Intake - Lean Pork (Active Comparator): Meal patterns will mimic a standard American diet (50% carbohydrate, 15% protein, 35% fat), providing an isonitrogenous 0.8 g/kg/d protein, and meeting individual estimated daily energy requirements. We have chosen 0.8 g/kg/d as it is the recommend dietary allowance for protein in the US. This arm's protein source will be from lean pork.
  Interventions: Other: Lean Pork vs Plant-Based Protein
- Low Quality Protein Intake - Plant-Based (Active Comparator): Meal patterns will mimic a standard American diet (50% carbohydrate, 15% protein, 35% fat), providing an isonitrogenous 0.8 g/kg/d protein, and meeting individual estimated daily energy requirements. We have chosen 0.8 g/kg/d as it is the recommend dietary allowance for protein in the US. This arm's protein source will be from plant-based protein (ie impossible burger, black bean burger, soy, etc).
  Interventions: Other: Lean Pork vs Plant-Based Protein

INTERVENTIONS:
Other: Lean Pork vs Plant-Based Protein — Participants will eat prepared study meals for three days that have either protein sourced from lean pork or plant-based sources.

SUMMARY:
We will be directly comparing a high-quality protein diet composed primarily of lean pork loin (PORK) to a lower-quality plant-based protein diet (PLANT) in individuals with prediabetes on muscle and whole-body protein turnover and glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females ages 40-65 years.
* 2. BMI 25 to ≤40 kg/m2 (or body fat % ≥25% in males or ≥36% in females)
* 3. Capable of providing informed consent.
* 4. COVID-19 negative and/or asymptomatic.
* 5. Willing to abstain from drinking alcohol or consuming marijuana and CBD products during the 4-day study meal period
* 6. HbA1c: 5.7-6.4% or fasting glucose 100-125 mg/dL

Exclusion Criteria:

* 1. Participant who does not/will not eat animal protein sources.
* 2. Allergy to wheat, soy, or common ingredients in plant-based protein products.
* 3. Body mass index <25 kg/m2 or >40 kg/m2.
* 4. Hemoglobin <10g/dL at screening.
* 5. Platelets <150,000/uL at screening.
* 6. History of chemotherapy or radiation therapy for cancer in the 6 months prior to enrollment.
* 7. History of gastrointestinal bypass/reduction surgery.
* 8. Pregnant or lactating individuals.
* 9. History of a chronic inflammatory disease (e.g. Lupus, Crohn's disease)
* 10. Currently receiving androgen (e.g., testosterone) or anabolic (e.g., GH, IGF-I) therapy.
* 11. Currently using prescription blood thinning medications.
* 12. Currently using corticosteroid medications (cortisone, hydrocortisone, prednisone, etc.).
* 13. Unable or unwilling to suspend aspirin use for 7 days prior to Visit 3 and Visit 7.
* 14. Unwilling to avoid using protein or amino-acid supplements during participation.
* 15. Unwilling to fast overnight.
* 16. Unwilling to avoid alcohol, marijuana and CBD products for the four study days.
* 17. Participants on glucagon-like-peptide-1 receptor agonist (GLP-1-RA) medications for <1 month or with less than one treatment dose (injection) every two weeks

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 24 hours
  Mixed muscle protein synthesis expressed as the fractional synthetic rate.
Whole Body Protein Balance | 24 hours
  Amount of net protein gained per unit of time.

SECONDARY OUTCOMES:
Whole Body Protein Synthesis | 24 hours
  Amount of protein produced per unit of time.
24-hour Mean Glucose | 24 hours
  Derived from continous glucose monitor data.

OTHER OUTCOMES:
Whole Body Protein Breakdown | 24 hours
  Amount of protein broken down per unit of time.
Whole Body Protein Flux | 24 hours
  Amount of protein turnover per unit of time.
Glucose Regulation and Homeostasis | 24 hours
  Derived from continuous glucose monitor data.

CONTACTS AND LOCATIONS:
Overall Officials: David Church, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No